CLINICAL TRIAL: NCT03243682
Title: The Alternating Bidirectional Versus The Standard Approach During Shock Wave Lithotripsy For Renal And Upper Lumbar Ureteric Stones. A Randomized Clinical Trial
Brief Title: The Alternating Bidirectional Versus The Standard Approach During Shock Wave Lithotripsy For Renal And Upper Lumbar Ureteric Stones
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Mahamed Hegazy, MD, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Bidirectional SWL
Record Dates: First submitted 2017-07-29; First posted 2017-08-09 (Actual); Last update posted 2017-08-09 (Actual); Status verified 2017-07

CONDITIONS: Urologic Diseases; Stones, Kidney; Stone, Urinary; Shock Wave Lithotripsy
Keywords: Shock wave lithotripsy; Bidirectional; Stones
MeSH Terms: conditions — Urologic Diseases; Kidney Calculi; Urinary Calculi; Calculi

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Bidirectional Shock Wave Lithotripsy (Active Comparator): alternating bidirectional (under and over table) approach
  Interventions: Procedure: Bidirectional Shock Wave Lithotripsy
- Standard Shock Wave Lithotripsy (Active Comparator): standard unidirectional approach
  Interventions: Procedure: Standard Shock Wave Lithotripsy

INTERVENTIONS:
Procedure: Bidirectional Shock Wave Lithotripsy — the alternating bidirectional (under and over table) approach during SWL for renal and upper lumbar ureteric stones
  Other Names: Bidirectional SWL
  Arms: Bidirectional Shock Wave Lithotripsy
Procedure: Standard Shock Wave Lithotripsy — the standard unidirectional approach during SWL for renal and upper lumbar ureteric stones
  Other Names: Standard SWL
  Arms: Standard Shock Wave Lithotripsy

SUMMARY:
compare the outcomes of SWL for renal and upper lumbar ureteric stones using the alternating bidirectional approach versus the standard approach.

DETAILED DESCRIPTION:
Shock wave lithotripsy (SWL) has been considered the preferred method for treating upper urinary tract stones since 1980s due to its minimally invasive characters and low morbidity. The overall stone free rates have been reported to be 80% to 90% .

In the presence of pregnancy, untreated urinary tract infection, decompensated coagulopathy, uncontrolled arrhythmia and abdominal aortic aneurysm, other treatment methods should be considered .

SWL is associated with some complications. The most common complications of SWL are renal colic (40%), gross hematuria (32%), urinary obstruction (30.9%), symptomatic bacteriuria (9.7%) and perirenal hematoma or subclinical subcapsular hematoma (4.6%).

There are many factors affecting the success of SWL as patient age, sex, body mass index (BMI), stone size, site and number, radiological renal features, congenital renal anomalies and presence of double-J (DJ) ureteric stent .

Regarding the renal stones, stones smaller than 10 mm had a success rate of 90%, while those larger than 10 mm had a success rate of 70%. Stones located in the renal pelvis and upper pole had a success rate of 87.3 and 88.5% respectively, while those located in the lower pole had a success rate of 69.5%. A single renal stone had a 78.3% success rate compared to 62.8% in multiple renal stones . Regarding the ureteric stones, stone size more than 10 mm was one of the strongest independent predictors of failure of SWL

Patients appear to have the best chance for successful SWL when they have small BMI and their stones are single and located in the renal pelvis . Skin to stone distance (SSD) measured by non-contrast computerized tomography scan (NCCT) has a significant role in the treatment of renal stones using SWL. Slow shock wave rate (60/min) is associated with increase in the success rate and decrease in pain, complication and number of session to achieve success when compared to rapid shock wave rate (120/min)

Some techniques were developed to increase the efficacy of SWL. In 1999, the bidirectional synchronous twin-pulse technique with variable angles between the shock wave reflectors was developed and it improved the quality and rate of stone disintegration in vitro and it was more effective than the traditional single generator and also it decreases the overall treatment times

The TWINHEADS 101 lithotripter comprises two identical under and over table reflectors to permit synchronous shock waves emission from two perpendicular directions to the same focal point. This technique intensifies and localizes the cavitations effects by the interacting focal zones of both reflectors, resulting in a better quality and rate of stone disintegration, especially with a right angle between the axes of the reflectors.

The first prospective clinical study was done in 2005 regarding synchronous twin-pulse SWL and it seems safe and effective for treating patients with renal and upper ureteric stones. The stone-free rate was 74% after one session and 100% after two sessions within a month

Based on the principle of the TWINHEADS lithotripter, we will use Dornier Gemini lithotripter to emit the shock waves from two different directions to the same focal point asynchronously for renal and upper lumbar ureteric stones.

ELIGIBILITY:
Inclusion Criteria:

* Patient criteria:

  1. Ability to give informed consent.
  2. Normal laboratory profile as regarding serum creatinine, liver function, platelets count and prothrombin time.
* Stone criteria:

  1. Single renal stone less than two cm or upper lumbar ureteric stone less than one cm.
  2. Radio-opaque stones.

Exclusion Criteria:

1. Bleeding tendency.
2. Poor kidney function.
3. Pregnancy.
4. Abdominal aortic aneurysm.
5. Indwelling DJ ureteric stent or percutaneous nephrostomy tube (PCN).
6. Congenital anomalies of the urinary tract.
7. Untreated urinary tract infection.
8. Obstructed urinary tract distal to the stone.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2016-09-01 (Actual); Primary Completion 2018-03-01 (Estimated); Study Completion 2018-03-01 (Estimated)

PRIMARY OUTCOMES:
stone free rate three months after the last session | 18 months
  residual less than 4 mm by non-contrast computerized tomography scan (NCCT)

SECONDARY OUTCOMES:
severity of complications after SWL in both groups | 18 months
  Clavien-Dindo scale of surgical complications

CONTACTS AND LOCATIONS:
Locations (1):
- Urology and Nephrology center, Al Mansurah, Egypt

REFERENCES:
- [Derived] Hegazy M, El-Assmy A, Ali-El-Dein B, Sheir KZ. The alternating bidirectional versus the standard approach during shock wave lithotripsy for upper lumbar ureteric stones: a randomized controlled trial. World J Urol. 2021 Jan;39(1):247-253. doi: 10.1007/s00345-020-03148-5. Epub 2020 Mar 23. PMID 32206888